CLINICAL TRIAL: NCT00525408
Title: Open Label, Randomized Multicentric Phase II Clinical Trial of Mycobacterium w in Combination With Docetaxel Versus Docetaxel in Metastatic Hormone Refractory Prostate Cancer.
Brief Title: A Study of Mycobacterium w Plus Docetaxel for Hormone Refractory Metastatic Prostate Cancer
Acronym: HRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Analysis report indicates trial futility
Sponsor: Cadila Pharnmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-60/1260
Record Dates: First submitted 2007-09-01; First posted 2007-09-05 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: HRPC; Metastatic Hormone Refractory Prostate Cancer; Docetaxel; Mycobacterium w
MeSH Terms: interventions — Mycobacterium w vaccine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Docetaxel+Mw
  Interventions: Biological: Mycobacterium w.
- 1 (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Mycobacterium w. — Immunomodulator
  Arms: 2
Drug: Docetaxel — Chemotherapeutic agent
  Arms: 1

SUMMARY:
This study proposed the comparison the overall survival, hematological toxicity, pain reduction score,PSA levels, tumor response, quality of life in two arms of HRPC patients from different parts of India.

DETAILED DESCRIPTION:
Prostate Cancer is a common health issue facing men worldwide in most of the patients cancer will shrink with hormonal therapy. In some cases cancer returns or continues to grow despite very low levels of circulating male hormones, which is called Androgen-Independent Prostate Cancer (AIPC) or Hormone Refractory Prostate Cancer (HRPC). Mycobacterium w is known to share multiple antigen including PSA. It administration is associated with antigen specific generation of cell mediated immunity. Docetaxel is found to useful in management of metastatic hormone refractory prostate cancer, which is associated with improved survival, tumor progression free survival with reduction in pain, serum PSA and improvement in quality of life. Cyclophosphamide 300mg/sq.m will be used to eliminate T-regulatory cell responsible immuno suppression. The vaccine Mycobacterium w will be administered on a day following cyclophosphamide. For better initiation of immune responses Docetaxel will be given seven days following first dose of Mycobacterium w.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate with clinical or radiologic evidence of metastatic disease.
* Disease progression during antiandrogen therapy, having surgical or medical castration status.
* Karnofsky Performance Status 50-100
* Normal cardiac function
* Life expectancy at least 24 weeks.
* Laboratory criteria for eligibility will include
* A neutrophil count of at least 1500 per cubic millimeter
* A hemoglobin level of at least 9 gm%
* A platelet count of at least 1000,000 per cubic millimeter.
* A total bilirubin not grater than 1.5 times the upper limit of the normal range for each institution.
* Serum creatinine levels not more than 1.5 times the upper limit of the normal range
* Written informed consent

Exclusion Criteria:

* Prior treatment with cytotoxic agents or radioisotopes
* Estrogen use for at least three months
* History of another cancer within the preceding five years (except basal or squamous-cell skin cancer)
* Brain or leptomeningeal metastases
* Symptomatic peripheral neuropathy of grade 2 or higher
* Uncontrolled intercurrent illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Median Survival time | 12 months
Time to Tumor Progression | 12 Months

SECONDARY OUTCOMES:
hematological toxicity, PSA levels, Quality of Life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir Rawal, MD, Principal Investigator — Rajiv Gandhi Cancer Institute; Arup Kumar Mandal, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Devakar Dalela, MD, Principal Investigator — Chatrapati Sahuji Mahraj Medical University; N K Mohanty, M.D., Principal Investigator — Safdarjang Hospital; Jayesh Dhabalia, MD, Principal Investigator — SEth G S Medical College & KEM Hospital; Arun Chawla, MD, Principal Investigator — Kasturba Medical College; Sujata Patwardhan, MD, Principal Investigator — LTMMC & LTMGH; P G Jayaprakash, MD, Principal Investigator — RCC, Trivandrum; Amil Lal Bhat, MD, Principal Investigator — S.P. Medical College & A.G. Hospitals; Raju T Chacko, MD, Principal Investigator — Christian Medical College, Vellore, India; Sushil Bhatia, MD, Principal Investigator — Choithram Hospital & Research Centre; Kim Mammen, MD, Principal Investigator — Christian Medical College, Ludhiana; K C Lakshmaiah, MD, Principal Investigator — Kidwai Memorial Istitute of Oncology; Rajeev Gupta, MD, Principal Investigator — Patel Hospital Pvt. Ltd.
Locations (14):
- India (14):
  - Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Kasturba Hospital,, Manipal, Karnataka
  - Regional Cancer Centre, Trivandrum, Kerala
  - Choithram Hospital & Research Centre, Indore, Madhya Pradesh
  - Seth G.S. Medical College & KEM Hospital, Pārel, Mumbai
  - Lokmanya Tilak Municipal Medical College & General Hospital, Sion, Mumbai
  - V.M. Medical College & Safdarjang Hospital, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute & Research Center, Rohini, National Capital Territory of Delhi
  - Patel Hospital Pvt. Ltd., Jalandhar, Punjab
  - Christian Medical College, Ludhiana, Ludhiana, Punjab
  - S.P. Medical College & A. G. of Hospitals, Bikaner, Rajashthan
  - Christian Medical College, Vellore, Tamil Nadu
  - Chatrapati Sahuji Mahraj Medical University, Lucknow, Uttar Pradesh